CLINICAL TRIAL: NCT05520164
Title: Effect of Maternal Heart Sound on Crying Time and Pain Level in Newborns During Heel Blood Collection: A Randomized Controlled Study
Brief Title: Effect of Maternal Heart Sound on Crying Time and Pain Level in Newborns During Heel Blood Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Pendik District Health Directorate (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Saglik Bilimleri U
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Pain; Infant, Newborn, Disease
Keywords: Pain; Newborn; Non-Drug Pain Management
MeSH Terms: conditions — Pain; Disease

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: The two separate clinicians conducting the assessment were masked to allow for impartiality.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Routine heel blood was taken from the control group. At the same time, the behaviors of newborns were recorded on camera throughout the procedure. At the end of the study, the camera recording was watched and scored by two midwives who had training in the Neonatal Pain Scale.
- Experimental Group (Experimental): The newborns in the experimental group listened to the recorded heart sounds of their mothers for 1 minute before the heel blood procedure, during the procedure and for 1 minute after the procedure. At the same time, the behaviors of newborns were recorded on camera throughout the procedure. At the end of the study, the camera recording was monitored and scored by two midwives trained in the Neonatal Pain Scale.
  Interventions: Other: Listening the maternal heart sound during the invasive interventions

INTERVENTIONS:
Other: Listening the maternal heart sound during the invasive interventions — Heart sounds of the newborns' own mothers were recorded on the voice recorder with the help of a hand doppler device. This sound was listened by the newborns in the experimental group during the heel blood procedure.
  Arms: Experimental Group

SUMMARY:
This study was carried out to determine the effect of maternal heart sound listened to by newborns during heel blood collection on pain level and crying time.

DETAILED DESCRIPTION:
The randomized controlled and experimental study was conducted with 60 newborns applied to a public family health center for heel blood collection. The infants in the experimental group (n=30) were listened to the maternal heart sound before, during, and after the heel blood collection procedure, and routine blood collection was applied to the control group (n=30). Newborn Information Form and Newborn Infant Pain Scale (NIPS) were used to collect data.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 38-41 weeks,
* Chronological age of 2-28 days,
* Without any physical, metabolic or genetic disease,
* Newborns who did not use any analgesic drugs before the procedure

Exclusion Criteria:

* Newborns whose heel blood cannot be taken at once

Ages: 2 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
The Newborn Infant Pain Scale (NIPS) | 15 minutes
  The Newborn Infant Pain Scale (NIPS) was used. NIPS: Scale Lawrence et al. (1993) was developed to evaluate the behavioral and physiological pain responses of preterm and term infants. The scale consists of five behavioral factors (facial expression, crying, arousal, arm and leg movements) and one physiological (breathing pattern) factor. The crying factor is given 0-1-2 points, the other factors are given 0-1 points, and the total score is between 0-7. A high score indicates greater severity of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye KOSE, Phd Student, Principal Investigator — Pendik District Health Directorate; Besey OREN, Associate Prof, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Pendik Mehmet Oguz Family Health Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Effect of interactive distraction versus cutaneous stimulation for venipuncture pain relief in school age children. — https://doi.org/10.5430/jnep.v5n4p32
- See also: Effect of inhalation aromatherapy with lavender essence on pain associated with intravenous catheter insertion in preschool children: a quasi-experimental study. Com — https://doi.org/10.1016/j.ctcp.2017.05.008